CLINICAL TRIAL: NCT00175825
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, 4 Parallel Groups, Dose-ranging Trial Evaluating the Efficacy and Safety of Brivaracetam Used as Adjunctive Treatment at Doses of 5, 20 and 50 mg/Day in b.i.d. Administration (Oral Tablets of 2.5 or 10 mg) for a Maximum of 7 Weeks in Subjects From 16 to 65 Years With Refractory Epilepsy Suffering From Partial Onset Seizures Whether or Not Secondarily Generalized
Brief Title: A Dose-ranging Study With Brivaracetam in Patients From 16 to 65 Years With Refractory Partial Onset Seizures.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01193
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Epilepsy
Keywords: Epilepsy: partial onset seizures; brivaracetam
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Matching Placebo tablets administered twice a day
  Interventions: Other: Placebo
- Brivaracetam 5 mg/day (Experimental): Brivaracetam 5 mg/day, 2.5 mg administered twice a day
  Interventions: Drug: Brivaracetam
- Brivaracetam 20 mg/day (Experimental): Brivaracetam 20 mg/day, 10 mg administered twice a day
  Interventions: Drug: Brivaracetam
- Brivaracetam 50 mg/day (Experimental): Brivaracetam 50 mg/day, 25 mg administered twice a day
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Other: Placebo — Daily oral dose of two equal intakes, morning and evening, of Placebo in a double-blinded way for the 7-week Treatment Period
  Arms: Placebo
Drug: Brivaracetam — Daily oral dose of two equal intakes, morning and evening, of Brivaracetam over the 7-week Treatment Period
  Other Names: Briviact
  Arms: Brivaracetam 20 mg/day; Brivaracetam 5 mg/day; Brivaracetam 50 mg/day

SUMMARY:
This trial will evaluate the efficacy and safety of brivaracetam (at doses of 5, 20 and 50 mg/day in twice a day administration) as add-on therapy in subjects with focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Male/female from 16 to 65 years
* Well-characterized focal epilepsy or epileptic syndrome according to the International League Against Epilepsy (ILAE) classification
* History of partial onset seizures
* Subjects having at least 4 partial onset seizures during the 4-week Baseline Period and at least 2 partial onset seizures during the 3 months prior to Visit 1
* Subjects taking 1 or 2 concomitant Antiepileptic drugs (AED(s)) that have been at a stable dose.

Exclusion Criteria:

* Seizure type IA non-motor as only seizure type
* Seizures occurring only in clusters
* Status epilepticus during the last 2 years before Visit 1
* History of cerebrovascular accident (CVA)
* Presence of any sign suggesting rapidly progressing brain disorder or brain tumor

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2005-11-07 (Actual); Primary Completion 2006-06-29 (Actual); Study Completion 2006-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (42):
- United States (26):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Fresno, California
  - Bradenton, Florida
  - Jacksonville, Florida
  - Chicago, Illinois
  - Paducah, Kentucky
  - Ruston, Louisiana
  - Bethesda, Maryland
  - Burlington, Massachusetts
  - Grand Rapids, Michigan
  - Rochester, Minnesota
  - Tupelo, Mississippi
  - Chesterfield, Missouri
  - Great Falls, Montana
  - Englewood Cliffs, New Jersey
  - Toms River, New Jersey
  - New York, New York
  - Wilmington, North Carolina
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Woonsocket, Rhode Island
  - Greenville, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
- Brazil (3):
  - Florianópolis
  - Salvador
  - São Paulo
- India (5):
  - Bangalore
  - Hyderabad
  - Lucknow
  - Parel Mumbai
  - Trivandrum
- Mexico (8):
  - Aguascalientes
  - Chichuahua
  - Chihuahua City
  - Guadalajara
  - Monterrey
  - San Luis Potosí City
  - Valle Oriente Garza Garcia
  - Zapopan

REFERENCES:
- [Result] Toledo M, Whitesides J, Schiemann J, Johnson ME, Eckhardt K, McDonough B, Borghs S, Kwan P. Safety, tolerability, and seizure control during long-term treatment with adjunctive brivaracetam for partial-onset seizures. Epilepsia. 2016 Jul;57(7):1139-51. doi: 10.1111/epi.13416. Epub 2016 Jun 6. PMID 27265725
- [Derived] Bresnahan R, Panebianco M, Marson AG. Brivaracetam add-on therapy for drug-resistant epilepsy. Cochrane Database Syst Rev. 2022 Mar 14;3(3):CD011501. doi: 10.1002/14651858.CD011501.pub3. PMID 35285519
- [Derived] Brandt C, Klein P, Badalamenti V, Gasalla T, Whitesides J. Safety and tolerability of adjunctive brivaracetam in epilepsy: In-depth pooled analysis. Epilepsy Behav. 2020 Feb;103(Pt A):106864. doi: 10.1016/j.yebeh.2019.106864. Epub 2020 Jan 12. PMID 31937513
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in November 2005 and concluded in June 2006.
Pre-assignment Details: Participant Flow refers to the Intention-to-treat (ITT) Set. 210 subjects were initially randomized, 2 subjects discontinued due to Lost to Follow-Up before first study drug intake.
Period: Overall Study
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Started | 54 | 50 | 52 | 52
Completed | 49 | 46 | 51 | 51
Not Completed | 5 | 4 | 1 | 1
Not completed — Adverse Event | 3 | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-to-Treat (ITT) Set.
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day | Total Title
Number analyzed (Participants) | 54 | 50 | 52 | 52 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 1 | 5 | 13
  Between 18 and 65 years | 51 | 46 | 50 | 47 | 194
  >=65 years | 0 | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.59 (11.26) | 32.72 (12.16) | 35.31 (13.66) | 30.92 (11.57) | 33.15 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 20 | 24 | 24 | 98
  Male | 24 | 30 | 28 | 28 | 110

OUTCOME MEASURES:

1. Secondary Outcome: Percentage Change From Baseline in Partial Onset Seizure Frequency Per Week (Type I) Over the 7-week Treatment Period
Description: Calculated as 7-day seizure frequency during the 7-week Treatment Period - 7-day seizure frequency during the Baseline Period, divided by the 7-day seizure frequency during the Baseline Period with this quantity multiplied by 100. A negative value in percent change from Baseline indicates a decrease in partial seizure frequency from Baseline.
Time Frame: Baseline, during the 7-week Treatment Period
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
percentage of change | -21.7 [-42.99 to 12.04] | -29.91 [-53.33 to -3.83] | -42.56 [-67.92 to 0.44] | -53.04 [-69.33 to -19.56]

2. Secondary Outcome: Seizure Frequency Per Week for All Seizures (Types I +II +III) Over the Treatment Period
Description: Types I+II+III seizure frequency (Type I: Partial (focal, local), Type II: Generalized (convulsive or nonconvulsive), Type III: Unclassified) per week will be derived from the seizure count information recorded on the daily record card (e.g. date, number, type of epileptic seizures) and is defined as the number of seizures standardized to a 7-day period.
Time Frame: During the 7-week Treatment Period
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
seizures per week
  Baseline | 2.23 [1.30 to 4.22] | 2.21 [1.38 to 5.00] | 2.50 [1.50 to 6.06] | 1.99 [1.36 to 3.97]
  Treatment | 1.81 [0.88 to 3.50] | 1.61 [0.75 to 4.34] | 1.70 [0.59 to 3.97] | 0.92 [0.69 to 2.05]

3. Secondary Outcome: Absolute Change From Baseline in Seizure Frequency Per Week for Partial Onset Seizures (Type I) Over the Treatment Period
Description: Calculated as 7-day Partial Onset Seizures (Type I) frequency during the 7-week Treatment Period 7-day seizure frequency during the Baseline Period. A negative value from Baseline indicates a decrease in partial seizure frequency from Baseline.
Time Frame: During the 7-week Treatment Period
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
seizures per week | -0.37 [-1.18 to 0.19] | -0.66 [-1.19 to -0.07] | -0.84 [-2.21 to -0.08] | -0.92 [-2.44 to -0.24]

4. Secondary Outcome: Absolute Change From Baseline in Seizure Frequency Per Week for All Seizures (Types I + II + III) Over the Treatment Period
Description: Calculated as 7-day seizure frequency during the 7-week Treatment Period 7-day seizure (Types I + II + III) frequency during the Baseline Period. A negative value from Baseline indicates a decrease in partial seizure frequency from Baseline.
Time Frame: During the 7-week Treatment Period
Measure: Median (Inter-Quartile Range); unit: seizures per week
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
seizures per week | -0.40 [-1.18 to 0.19] | -0.66 [-1.19 to -0.07] | -0.80 [-2.21 to -0.08] | -0.92 [-2.44 to -0.37]

5. Secondary Outcome: Percentage Change From Baseline in Seizure Frequency Per Week for All Seizures (Types I + II + III) Over the Treatment Period
Description: as for outcome 1
Time Frame: During the 7-week Treatment Period
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
percentage of change | -24.35 [-43.61 to 12.00] | -29.91 [-53.33 to -3.83] | -41.57 [-65.31 to 0.44] | -53.05 [-69.33 to -22.82]

6. Secondary Outcome: Responder Rate in Partial Onset Seizures (Type I) Over the Treatment Period
Description: A responder was defined as a subject with a >= 50 % reduction in seizure frequency per week from the Baseline Period to the end of the Treatment Period.
Time Frame: During the 7-week Treatment Period
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
percentage of participants | 16.7 | 32.0 | 44.2 | 55.8

7. Secondary Outcome: Percentage of Subjects With Categorized Response to the Treatment in Partial Onset Seizures (Type I) Over the Treatment Period
Description: Categories of percentage reductions in seizures from baseline were as following: < -25 %; -25 % to <25 %; 25 % to <75 %; 75 % to <100 %; 100 %.
Time Frame: During the 7-week Treatment Period
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
percentage of participants
  < -25% | 18.5 | 8.0 | 9.6 | 13.5
  -25% to <25% | 35.2 | 38.0 | 30.8 | 13.5
  25% to <75% | 40.7 | 42.0 | 40.4 | 55.8
  75% to <100% | 1.9 | 4.0 | 11.5 | 9.6
  100% | 3.7 | 8.0 | 7.7 | 7.7

8. Secondary Outcome: Percentage of Subjects Who Are Seizure Free During the 7-week Treatment Period
Description: A subject was considered seizure free, if no seizure was reported during the 7-week Treatment Period.
Time Frame: During the 7-week Treatment Period
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
percentage of participants
  Completed the Period | 1.9 | 8.0 | 7.7 | 5.8
  Discontinued from the Period | 1.9 | 0 | 0 | 0

9. Secondary Outcome: Number of Seizure-free Days Per 4 Weeks
Description: A day was considered seizure-free, if no seizure was reported during 24 hours.
Time Frame: Baseline, during the 7-week Treatment Period
Measure: Median (Inter-Quartile Range); unit: Days/4 Weeks
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
Days/4 Weeks | 22.66 [16.57 to 24.57] | 22.86 [15.43 to 25.14] | 22.84 [18.57 to 25.71] | 24.65 [21.14 to 25.86]

10. Secondary Outcome: Time to Nth (n= 1, 5, 10) Seizure During the 7-week Treatment Period
Description: Number of days to first, fifth, and tenth seizure after baseline.
Time Frame: During the 7-week Treatment Period
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
days
  Number of days to first seizure after baseline | 4.0 [3.0 to 6.0] | 4.0 [3.0 to 7.0] | 4.5 [2.0 to 8.0] | 7.0 [4.0 to 13.0]
  Number of days to fifth seizure after baseline | 17.0 [13.0 to 22.0] | 20.0 [17.0 to 27.0] | 18.5 [14.0 to 29.0] | 32.5 [23.0 to 42.0]
  Number of days to tenth seizure after baseline | 32.0 [23.0 to 45.0] | 38.0 [27.0 to NA] — upper limit is not available | 39.0 [23.0 to NA] — upper limit is not available | 57.0 [49.0 to NA] — upper limit is not available

11. Primary Outcome: Partial Onset Seizure Frequency Per Week During the 7-week Treatment Period
Description: Calculated as 7-day partial onset seizure frequency.
Time Frame: During the 7-week Treatment Period
Measure: Median (Inter-Quartile Range); unit: Seizures per week
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
Number analyzed (Participants) | 54 | 50 | 52 | 52
Seizures per week | 1.81 [0.88 to 3.50] | 1.61 [0.75 to 4.34] | 1.55 [0.57 to 3.83] | 0.92 [0.69 to 2.05]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 5 mg/Day; ANCOVA with baseline seizure frequency per week and each of the stratification factors as independent variables; Test type: Superiority or Other; p = 0.240, ANCOVA; Percent reduction over Placebo = 9.8, 95% CI 2-sided [-7.2 to 24.0]
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 20 mg/Day; ANCOVA with baseline seizure frequency per week and each of the stratification factors as independent variables; Test type: Superiority or Other; p = 0.062, ANCOVA; Percent reduction over Placebo = 14.9, 95% CI 2-sided [-0.8 to 28.2]
Statistical Analysis 3: Comparison: Placebo vs Brivaracetam 50 mg/Day; ANCOVA with baseline seizure frequency per week and each of the stratification factors as independent variables; Test type: Superiority or Other; p = 0.004, ANCOVA; Percent reduction over Placebo = 22.1, 95% CI 2-sided [7.6 to 34.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline until Safety Visit (up to 3 months).
Description: Adverse Events refer to the Safety Population consisting of all subjects who were dispensed medication.
Arm/Group | Placebo | Brivaracetam 5 mg/Day | Brivaracetam 20 mg/Day | Brivaracetam 50 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/50 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/50 | 1/52 | 0/52
Other Adverse Events (participants affected / at risk) | 15/54 | 13/50 | 8/52 | 10/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Brivaracetam 5 mg/Day (N=50) | Brivaracetam 20 mg/Day (N=52) | Brivaracetam 50 mg/Day (N=52)
Neurotoxicity (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Brivaracetam 5 mg/Day (N=50) | Brivaracetam 20 mg/Day (N=52) | Brivaracetam 50 mg/Day (N=52)
Neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 1
Fatigue (General disorders) | 2 | 0 | 2 | 3
Influenza (Infections and infestations) | 4 | 4 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 4
Headache (Nervous system disorders) | 4 | 4 | 2 | 1
Somnolence (Nervous system disorders) | 4 | 1 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days